CLINICAL TRIAL: NCT04935918
Title: PROSPECTIVE STUDY EVALUATING THE SAFETY AND EFFECTIVENESS OF ADJUSTABLE CONTINENCE THERAPY (ACT) BALLOONS FOR THE MANAGEMENT OF URINARY INCONTINENCE IN CHILDREN WITH BLADDER EXSTROPHY OR INCONTINENT EPISPADIAS
Brief Title: EVALUATION OF THE SAFETY AND EFFICACY OF ADJUSTABLE CONTINENCE THERAPY BALLOONS IN BLADDER EXSTROPHY AND INCONTINENT EPISPADIAS PATIENTS
Acronym: ACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-41
Record Dates: First submitted 2021-06-08; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Bladder Exstrophy
MeSH Terms: conditions — Bladder Exstrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm 1 (Experimental): Children with bladder exstrophy or isolated epispadias
  Interventions: Device: ACT

INTERVENTIONS:
Device: ACT — Implantation of ACT balloon, Uromedica (Irvine, CA, USA) periurethrally at the bladder neck. The ACT system is a permanent implant designed for the correction of incontinence in patients.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of a minimally invasive surgical procedure with ACT (Adjustable Continence Therapy) balloons implantation for the treatment of urinary incontinence in children with bladder exstrophy or isolated epispadias.

The ACT therapy consists of two small adjustable silicone balloons connected with a tubing to a port, surgically placed around the bladder neck, one on each side of the urethra.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls > 5 years with bladder exstrophy or isolated epispadias;
* sphincteric incontinence (leak point pressure < 45 cm d'H20, open bladder neck during filling, stress urinary incontinence);
* normal renal function (eGFR > 90ml/min);
* no (or stable) upper urinary tract dilatation in ultrasound.

Exclusion Criteria:

* under 5 years or more than 18 years old;
* renal insufficiency (acute or chronic);
* evolutive deterioration of the upper urinary tract (hydronephrosis);
* unmanageable detrusor instability;
* residual volume greater than 100 ml after voiding;
* bleeding disorders.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the clinical impact of ACT balloon on urinary continence with pad weight | 24 months
  Therapeutic success will be based on whether patients demonstrate at least a 50% reduction in 24 hour Pad weight at 6, 12 and 24 months follow-up compared to the pad weight results at baseline.

SECONDARY OUTCOMES:
Number of pads per day (voiding diary) | 6, 12 and 24 months
  Change of number of peds changed per day from baseline to 6, 12 and 24 months (the best : 0 pads changed a day).
Number of incontinence episodes per day (voiding diary) | 6, 12 and 24 months
  Change in number of incontinence episodes per day from baseline to 6, 12 and 24 months (the best : 0)
PIN-Q questionnaire | 6, 12 and 24 months
  Change on validated incontinence quality of life questionnaire from baseline to 6, 12 and 24 months
Incidence of urethral stricture and device erosion after ACT implantation | 6, 12 and 24 months
  Cumulative incidence of ACT related clinically relevant urethral structure and device erosions (the best : 0)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO-PRADALIE, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, PACA, France